CLINICAL TRIAL: NCT01030263
Title: A Prospective Randomized Trial Comparing Yield of Confocal Endomicroscopy Guided Biopsies With Random Biopsies in the Detection of Specialized Columnar Epithelium in Barrett's Esophagus
Brief Title: A Trial Comparing Yield of Confocal Endomicroscopy Guided Biopsies
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The investigators left the institution.
Sponsor: Mayo Clinic (Other)
Responsible Party: Ananya Das MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-001090
Record Dates: First submitted 2009-12-07; First posted 2009-12-11 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-03

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CEM (Experimental): Biopsies obtained with fluorescence-aided confocal endomicroscopy.
  Interventions: Other: Fluorescence-aided confocal endomicroscopy guided biopsy.
- RFQ (Other): Random four-quadrant biopsies.
  Interventions: Other: Random four-quadrant biopsies.

INTERVENTIONS:
Other: Fluorescence-aided confocal endomicroscopy guided biopsy. — Fluorescence-aided confocal endomicroscopy guided biopsy.
  Arms: CEM
Other: Random four-quadrant biopsies. — Random four-quadrant biopsies.
  Arms: RFQ

SUMMARY:
We wish to determine whether biopsies obtained with the technique of fluorescence-aided confocal endomicroscopy will detect more patients with specialized columnar epithelium than random biopsies among patients with Barrett's esophagus who are being monitored with endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18.
* Barrett's esophagus
* Acid suppressive therapy
* Endoscopic surveillance

Exclusion Criteria:

* Pregnancy or lactation
* Allergy to fluorescein
* Endoscopic esophagitis Los Angeles classification A to D
* Mucosal irregularity or nodules suspicious for dysplastic or cancerous lesion
* Obvious mass lesions or cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Whether specialized columnar epithelium was detected. | At biopsy on Day 0.

CONTACTS AND LOCATIONS:
Overall Officials: Ananya Das, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States